CLINICAL TRIAL: NCT02308852
Title: Improving Bi-manual Activities in Stroke Patients With Application of Neuro-stimulation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Professer Yves Vandermeeren, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B039201317382
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Stroke; Deficit in Manual Activities
Keywords: bi-manual , motor skill learning , stroke , chronic patients,neuro-rehabilitative robot
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: tDCS real versus sham tDCS (this is what this is)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- real tDCS (Active Comparator): Patients will receive non-invasive and painless brain stimulation over the brain areas involved in cognitive aptitudes.
  tDCS will be applied during 20 minutes while patients will perform motor bimanual tasks
  Interventions: Device: tDCS
- Sham tDCS (Placebo Comparator): this will be exactly as for "real tDCS" unless that the tDCS will be rapidly turned off, unbeknown from patients-therapist-examinator (double-blind trial)
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS

SUMMARY:
Noninvasive brain stimulations (NIBS) will be used in healthy volunteers and in chronic stroke patients to improve bimanual activities and motor learning.

Functional magnetic resonance imaging will be used to evaluate the mechanisms underlying bimanual activities and motor learning in healthy volunteers and in chronic stroke patients.

A neuro-rehabilitation robot (REA2PLAN, AXINESIS, Louvain-la-Neuve, Belgium) will be used for motor learning.

DETAILED DESCRIPTION:
tDCS will be used in a sham-controlled, double-blind, randomized, cross-over control trial in chronic stroke patients with motor deficits. After informed consent and recruitment, patients will be randomly (computer method) allocated to real or sham tDCS, that will be applied during performance of bimanual activities and/or motor learning. A few minutes/hours/days/weeks after completing one trial's arm, the patients will enter the other trial's arm (double-blind cross-over design).

Baseline and follow-up outcomes about bimanual and unimanual motor tasks will be collected.

For a subset of subjects, motor learning and data acquisition will be performed with a neuro-rehabilitation robot (REA2PLAN, AXINESIS, Louvain-la-Neuve, Belgium) .

ELIGIBILITY:
Inclusion Criteria:

• stroke with at least slight deficit

Exclusion Criteria:

* epilepsy
* contraindication to tDCS and/or to fMRI
* presence of metal in the head
* inability to understand / complete behavioral tasks
* chronic intake of alcohol or recreational drugs
* major health condition
* presence of pacemaker (for the fMRI part only)
* pregnancy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
bimanual coordination | up to 2 hours after intervention. Recall test at 1 week and up to,2,3,4 weeks after the intervention
  The effect of intervention on bimanual motor coordination will be quantified before, during and after executive tasks.

SECONDARY OUTCOMES:
standard unimanual evaluation | immediately, 30, 60 min; and up to 2 hours after intervention. Recall test at 1 week and up to,2,3,4 weeks after the intervention)
  Performance on motor skill learning tasks and on different commonly used tasks (Purdue Pegboard, hand dynamometer, pinch dynamometer, 9-HPT, motor skill learning with a videogame, ...) will be measured to explore the impact of tDCS on these parameters in chronic stroke patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital CHU Dinant Godinne UcL Namur, Yvoir, Belgium

REFERENCES:
- [Derived] De Laet C, Herman B, Riga A, Bihin B, Regnier M, Leeuwerck M, Raymackers JM, Vandermeeren Y. Bimanual motor skill learning after stroke: Combining robotics and anodal tDCS over the undamaged hemisphere: An exploratory study. Front Neurol. 2022 Aug 18;13:882225. doi: 10.3389/fneur.2022.882225. eCollection 2022. PMID 36061986
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411